CLINICAL TRIAL: NCT05064592
Title: Retrospective Study on Prolonged Sedation Effects With Inhaled Agents in Pediatric Intensive Care Unit
Brief Title: Retrospective Study on Prolonged Sedation Effects With Inhaled Agents in PICU
Acronym: RESPIRE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211236
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation
Keywords: Artificial ventilation; Pediatric intensive care unit; Prolonged sedation effects; Halogenated anesthetic gases; Inhaled agents; Benzodiazepines in combination with opioids; Halogenated anesthetic gases efficacity and tolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Medical records of minor patients hospitalized between 2015 and 2020 in PICU and having been under sedation and prolonged invasive mechanical ventilation (> 72h).

SUMMARY:
The objective of the study is to evaluate the effects of halogenated gases on sedation and analgesia, to describe the tolerance and to determine the risk factors for failure, in pediatric intensive care patients during prolonged sedation.

This study will be based on the medical records of patients hospitalized between 2015 and 2020.

DETAILED DESCRIPTION:
Sedation is a major therapeutic element in patients in intensive care under artificial ventilation, in order to allow their comfort and patient-ventilator synchronization. The use of benzodiazepines in combination with opioids is common practice. However, during prolonged sedation, the effects wane, then the doses must be increased, responsible for an increase in the incidence of a significant withdrawal syndrome in the recovery phase, a source of delay in extubation or early reintubation.

The use of halogenated anesthetic gases is now possible in pediatric intensive care in these patients on artificial ventilation.

Their efficacy and tolerance in prolonged use must be evaluated. Their use could improve the sedative effects, reduce the doses of benzodiazepines and opioids used, and reduce unwanted effects in terms of withdrawal syndrome.

The objective of the study is to evaluate the effects of halogenated gases on sedation and analgesia, to describe the tolerance and to determine the risk factors for failure, in pediatric intensive care patients during prolonged sedation.

This study will be based on the medical records of patients hospitalized between 2015 and 2020.

ELIGIBILITY:
Inclusion Criteria:

* Minor patient over 1 month old (and over 36 WA of corrected age) and under 18 years old
* Hospitalized in neonatal or pediatric intensive care unit
* Invasive mechanical ventilation over 72 hours
* Prolonged sedation greater than 72 hours

Exclusion Criteria:

- Opposition of the holders of parental authority of the minor patient or the adult patient to the use of the data for the study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Minor patients hospitalized between 2015 and 2020 in PICU and having been under sedation and prolonged invasive mechanical ventilation (> 72h).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Dosages of hypnotics first 24 hours following the introduction of halogens | Day 0
  Show a reduction in hypnotics dosages, calculated in Midazolam equivalent in µg / kg / h, during the first 24 hours after the introduction of halogens.
  A decrease will be significant if it is greater than 20% compared to the basal level before initiation of the halogens.

SECONDARY OUTCOMES:
Dosages of opioids in the 24 hours following the introduction of halogens | Day 0
  Show a reduction > 20% in opioids dosages (calculated in morphine equivalent, in µg / kg / h, in the 24 hours following the introduction of halogens.
Dosages of ketamine within 24 hours of the introduction of halogens | Day 0
  Show a reduction >20% in ketamine dosages within 24 hours of the introduction of halogens (mg / kg / h).
Morphinic / hypnotic dosages at the end of halogenated use | Day 0
  Show a reduction > 20% in morphinic / hypnotic dosages at the end of halogenated use (> 24 hours).
Clinical sedation score | Day 0
  COMFORT BEHAVIOUR scale. Measures pain and excess sedation in intensive care, starting in the neonatal period.
  Score: from 6 to 30 :
  Excess sedation: 6 to 10 Comfortable child, sedated without excess: 11 to 17 Child in borderline condition, possible pain: 17 to 22 Child clearly uncomfortable, painful: 23 to 30
Hypnotics / sedatives / curares dosages in populations of ARDS patients at the end of the use of halogens | Day 0
  Show a reduction> 20% in hypnotics / sedatives / curares dosages (µg/kg/h) in populations of Acute Respiratory Distress Syndrome patients (ARDS patients) with and without extracorporeal membrane oxygenation (ECMO) at the end of the use of halogens (> 24 hours).
Ventilatory parameters in patients with ARDS during the period of halogen use | Day 0
  Show a reduction > 20% in ventilatory parameters (PEEP in mmHg, Tidal volume in ml, PaO2/FiO2 ratio) in patients with ARDS during the period of halogen use (<24 hours).
Total duration of sedation, analgesia and curarization | Day 0
  Determine the total duration of sedation, analgesia and curarization.
Halogenated failure criteria | Day 0
  Comparison of patients who shown an improvement of the COMFORT B scale 24 hours after introducing halogenated between patients who shown no significant reduction of COMFORT B scale.
Withdrawal syndrome: morphine and hypnotics | Day 0
  Determine the proportion of withdrawal syndrome : morphine and hypnotics in %.
Tachyphylaxis to halogenated | Day 0
  Withdrawal syndrome within 24 hours of stopping halogenated: proportion of tachyphylaxis to halogenated.
Adverse effects of secondary to prolonged administration of Sevoflurane or Isoflurane | Day 0
  Describe the proportions of side effects: Malignant hyperthermia, Arterial hypotension, Tachycardia, Bradypnea or apnea, Bronchospasm, Arrhythmias, Cytolytic hepatitis, Chills, nausea, vomiting upon awakening, Irritation of the respiratory tract, Headache.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Louis Léger, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Léo Berger, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Armand Trousseau, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halogenated volatile anaesthetics for prolonged sedation in pediatric intensive care unit: first experience in two French pediatric intensive care units. https://doi.org/10.1007/s44253-023-00009-y.Léo Berger, Yohan Soreze, Jérome Rambaud, Julie Starck, Yael Levy, Pierre Tissières, Jordi Miatello, Luc Morin & Pierre-Louis Léger